CLINICAL TRIAL: NCT04901104
Title: Long-term Prognosis After Thymosin Alpha 1 Treatment in Patients With Sepsis: A Multicenter Cohort Study
Brief Title: Long-term Prognosis of Patients With Sepsis After Immunotherapy
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wu Jianfeng, chief physician, Sun Yat-sen University
Other Study IDs: Long-term prognosis in sepsis
Record Dates: First submitted 2021-05-24; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Long-term Effects of Thymosin Alpha 1 Treatment
Keywords: long-term; thymosin alpha 1; sepsis; immunotherapy
MeSH Terms: conditions — Sepsis | interventions — Thymalfasin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- thymosin α1 group: The patient was treated with thymosin α1 in sepsis
  Interventions: Drug: Thymosin Alpha1
- placebo group: The patient was treated without thymosin α1 in sepsis

INTERVENTIONS:
Drug: Thymosin Alpha1 — Drug interventions have been done in previous clinical studies
  Groups: thymosin α1 group

SUMMARY:
Current clinical studies of thymosin α1 for sepsis have focused on short-term outcomes (28-day or 90-day mortality), and lack of clinical data on long-term outcomes (3 year mortality) of patients with sepsis after immunotherapy.

Based on the preliminary clinical study (NCT02867267), this study will conduct long-term follow-up for sepsis patients to provide data support for the long-term prognosis of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis patients in the TESTS study Patients who discharged from hospital after recovery

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sepsis patients who discharged from hospital after recovery in the TESTS study
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
three years mortality | 3 years
  Mortality rate of patients treated with thymosin α1 or placebo within 3 years

SECONDARY OUTCOMES:
Recurrence rate of sepsis | 5 years
  Percentage of recurrent sepsis within 5 years of discharge sepsis patients
one year mortality | 1 year
  Mortality rate of patients treated with thymosin α1 or placebo within 1 year
Five years mortality | 5 years
  Mortality rate of patients treated with thymosin α1 or placebo within 5 years
short form 36 questionnaire | 1 year
  Quality of life of sepsis patients after 1 year of thymosin α1 or placebo treatment

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: This study is a follow-up study of TESTS study — http://clinicaltrials.gov/ct2/show/study/NCT02867267